CLINICAL TRIAL: NCT03908450
Title: Treatment of Coronary De-novo Stenosis by a Sirolimus Coated Balloon or a Paclitaxel Coated Balloon Catheter
Acronym: SCBDENOVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InnoRa GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SI-DN-01
Record Dates: First submitted 2019-04-02; First posted 2019-04-09 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Outcomes Assessor
Masking Description: angiographies blinded to treatment groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control intervention (Active Comparator): Predilatation of coronary de-novo stenosis followed by a SeQuent®Please or SeQuent®Please Neo balloon (paclitaxel 3.0 μg/mm²)
  Interventions: Device: PTCA of coronary de novo lesion PCB
- Experimental intervention (Experimental): Predilatation of coronary de-novo stenosis followed by a sirolimus coated SeQuent®SCB balloon (sirolimus 4.0 μg/mm²)
  Interventions: Device: PTCA of coronary de novo lesion SCB

INTERVENTIONS:
Device: PTCA of coronary de novo lesion PCB — PTCA of coronary de novo lesion with drug coated balloon
  Arms: Control intervention
Device: PTCA of coronary de novo lesion SCB — PTCA of coronary de novo lesion with drug coated balloon
  Arms: Experimental intervention

SUMMARY:
To examine the treatment of coronary de-novo stenosis with a sirolimus coated balloon versus a paclitaxel coated balloon

DETAILED DESCRIPTION:
To examine the treatment of coronary de-novo stenosis with a sirolimus coated balloon versus a paclitaxel coated balloon. Prospective, multicenter, randomized, single-blind, 70 patients. Experimental intervention: Predilatation of coronary de-novo stenosis followed by a sirolimus coated SeQuent®SCB balloon (sirolimus 4.0 μg/mm²). Control intervention: Predilatation of coronary de-novo stenosis followed by a SeQuent®Please or SeQuent®Please Neo balloon (paclitaxel 3.0 μg/mm²). Follow-up per patient: 30 days telephone call; 6 months angiographic + 12 months. clinical follow up

Key inclusion criteria: > 18 years of age, Clinical evidence of stable or unstable angina or a positive functional study, Patients with significant coronary de-novo stenosis (≥ 70% diameter stenosis or intermediate ≥ 50% to <70% diameter stenosis with positive functional test or symptom of ischemia), Successful lesion preparation (no flow-limiting dissection or a residual stenosis > 30%).

Key exclusion criteria: Acute myocardial infarction within the past 72 hours (STEMI or NSTEMI), Intolerance and / or allergy to Sirolimus, Intolerance or allergy to Paclitaxel and/or the delivery matrix (main ingredient: iopromide), Patients with an ejection fraction of < 30 %, Reference vessel diameter (RVD) < 2.5 mm, Contraindication for whichever necessary accompanying medication.

Primary efficacy endpoint: late lumen loss in-segment at 6 months. Key secondary endpoints: Procedural Success: < 30% final diameter stenosis, no flow-limiting dissection (type C or higher), TIMI III flow, and the absence of in-hospital MACE. MACE: cardiac death, target vessel myocardial infarction, and clinically driven target lesion revascularization in-hospital at 6 and at 12 months Individual clinical endpoints at 6 and at 12 months: cardiac death, target lesion myocardial infarction, clinically driven target lesion revascularization, (stenosis ≥ 50% at follow-up angiography)

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of stable or unstable angina or a positive functional study
* Patients with significant coronary de-novo stenosis (≥ 70% diameter stenosis or intermediate ≥ 50% to <70% diameter stenosis with positive functional test or symptom of ischemia)
* Successful lesion preparation (no flow-limiting dissection or a residual stenosis > 30%)

Exclusion Criteria:

* Acute myocardial infarction within the past 72 hours (STEMI or NSTEMI)
* Intolerance and / or allergy to Sirolimus
* Intolerance or allergy to Paclitaxel and/or the delivery matrix (main ingredient:

iopromide)

* Patients with an ejection fraction of < 30 %
* Reference vessel diameter (RVD) < 2.5 mm
* Contraindication for whichever necessary accompanying medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
late lumen loss in-segment | 6 months
  angiographic minimal lumen diameter in-segment at 6 months minus minimal lumen diameter at baseline

SECONDARY OUTCOMES:
Procedural Success | in hospital
  < 30% final diameter stenosis, no flow-limiting dissection (type C or higher), TIMI III flow, and the absence of in-hospital MACE
MACE MACE | at 6 and at 12 months
  cardiac death, target vessel myocardial infarction, and TLR target lesion revascularization in-hospital at 6 and at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Scheller, MD, Principal Investigator — Clinical and Experimental Interventional Cardiology, University of Saarland
Locations (4):
- Germany (3):
  - Klinik fuer Innere Medizin III, Universitaetsklinikum des Saarlandes, Homburg/Saar, Saarland
  - Herzzentrum Dresden, Universitätsklinik an der Technischen Universität Dresden, Dresden
  - Klinik für Innere Medizin III - Kardiologie Paul Gerhardt Stift, Wittenberg
- Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali RM, Abdul Kader MASK, Wan Ahmad WA, Ong TK, Liew HB, Omar AF, Mahmood Zuhdi AS, Nuruddin AA, Schnorr B, Scheller B. Treatment of Coronary Drug-Eluting Stent Restenosis by a Sirolimus- or Paclitaxel-Coated Balloon. JACC Cardiovasc Interv. 2019 Mar 25;12(6):558-566. doi: 10.1016/j.jcin.2018.11.040. PMID 30898253
- [Derived] Scheller B, Mangner N, Jeger RV, Afan S, Mahfoud F, Woitek FJ, Fahrni G, Schwenke C, Schnorr B, Kleber F. A randomised trial of sirolimus- versus paclitaxel-coated balloons for de novo coronary lesions. EuroIntervention. 2024 Nov 4;20(21):e1322-e1329. doi: 10.4244/EIJ-D-23-00868. PMID 39492703